CLINICAL TRIAL: NCT07333781
Title: Effects of a Communication Skills Training Program for Occupational Therapy Interns in Mental Health
Brief Title: Effects of Communication Training for Mental Health Occupational Therapy Interns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202200268B0
Record Dates: First submitted 2025-12-24; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2022-07

CONDITIONS: Communication
Keywords: communication skills; communication skills training; occupational therapy
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: Intervention group receives the iCOT program; comparison group uses historical active control data.
Who Masked: Outcomes Assessor
Masking Description: Single-blind. Expert raters evaluating communication skills are blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCOT Communication Training (Experimental): Participants receive the iCOT (Intervention Protocol for Communication Skills of Occupational Therapy Interns) communication skills training program. The program includes structured instructional content based on therapist-patient communication models, teaching strategies designed for OT interns, and a training sequence integrated into internship schedules. Training is delivered during the internship period.
  Interventions: Behavioral: iCOT
- Active Control (Historical Data) (Active Comparator): This arm uses historical data from a previous cohort of occupational therapy interns, clinical supervisors, and patients. The cohort includes 44 interns, 9 supervisors, and 97 patients who completed standard internship training without the iCOT program. Their communication performance, measured with the Gap-Kalamazoo Communication Skills Assessment Form (GKCSAF), serves as the comparison group.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: iCOT — The intervention group receives the iCOT program, which includes:
  1. Online training through Moodle with instructional videos, expert demonstrations, and scenario-based quizzes requiring full completion; and
  2. Multi-source feedback from patients, clinical supervisors, and experts using structured communication assessment tools. The program aims to improve communication skills during mental health clinical practice.
  Other Names: An intervention protocol for communication skills of occupational therapy interns in in the field of mental health clinical practice
  Arms: iCOT Communication Training
Behavioral: Active Control — The active control group receives the standard communication training used in routine internship education. Interns complete three recorded patient interviews during the internship, followed by supervisor feedback using the GKCSAF. The control group does not receive the iCOT online modules, expert demonstrations, scenario-based training, or patient feedback. Total training time is approximately 2.5 hours shorter than the intervention group.
  Other Names: Standard Communication Training
  Arms: Active Control (Historical Data)

SUMMARY:
The goal of this clinical trial is to develop and test a new communication skills training program for occupational therapy (OT) interns in mental health practice, called the Intervention Protocol for Communication Skills of Occupational Therapy Interns (iCOT). The main questions are:

Does iCOT improve interns' communication skills in the short term?

The study has two parts. First, researchers will develop the iCOT program using expert input, feedback from recent graduates, and feasibility testing with interns, supervisors, and patients. Second, the study will test iCOT using a single-blind design. Expert raters, who do not know which group each intern belongs to, will evaluate communication skills using the Gap-Kalamazoo Communication Skills Assessment Form (GKCSAF).

The intervention group will receive iCOT training. The comparison group will use data from a previous study of interns, supervisors, and patients. Communication skills will be rated by experts (primary outcome) and by supervisors, patients, and interns (secondary outcomes).

DETAILED DESCRIPTION:
Communication skills are essential for occupational therapy (OT) practitioners working in mental health settings. Strong communication skills improve treatment quality, therapeutic relationships, and clinical outcomes. However, there is currently no evidence-based communication training specifically designed for OT interns in mental health. This gap limits both clinical education and research in the field.

This study aims to develop and evaluate a structured communication skills training program for mental-health OT interns, called the Intervention Protocol for Communication Skills of Occupational Therapy Interns (iCOT). The study has two phases and uses a single-blind clinical trial design, in which expert raters are blinded to group assignment.

Phase 1: Development of the iCOT Program

In Phase 1, researchers will create the iCOT training program through several steps:

Teaching content: Materials will be designed based on established models of therapist-patient communication in mental health.

Teaching methods: Instructional strategies will be developed to fit OT interns' learning needs.

Procedure design: The training sequence will align with internship schedules and clinical workflow.

Expert validation: Three clinical experts, two university instructors, and five recent graduates will review and validate the initial version.

Feasibility testing: Five interns, their clinical supervisors, and patients will pilot-test the program to refine the final version.

Phase 2: Evaluation of iCOT Effectiveness

In Phase 2, the finalized iCOT program will be tested. The intervention group will include OT interns, clinical supervisors, and patients participating in the current study. The comparison group will consist of previously collected data from 44 interns, 9 supervisors, and 97 patients.

The primary outcome is interns' communication performance evaluated by blinded expert raters using the Gap-Kalamazoo Communication Skills Assessment Form (GKCSAF). Secondary outcomes include GKCSAF ratings completed by clinical supervisors, patients, and the interns themselves.

This study will provide the first evidence-based communication skills training protocol tailored to OT interns in mental health and may support future improvements in clinical education and quality of care.

ELIGIBILITY:
Inclusion Criteria:

Occupational therapy interns: willing to participate; no additional inclusion or exclusion criteria.

Clinical supervisors (occupational therapists): willing to participate; no additional inclusion or exclusion criteria.

Patients:

Diagnosed with any DSM-5 mental disorder

Age 20 years or older

Able to provide informed consent

Adequate verbal communication ability

Exclusion Criteria:

Patients: severe cognitive impairment (e.g., aphasia or inability to follow three-step commands).

Interns and supervisors: none.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Expert-rated communication skills performance | Baseline and immediately after completion of the intervention.
  Blinded expert raters evaluate interns' communication skills using the Gap-Kalamazoo Communication Skills Assessment Form (GKCSAF).

SECONDARY OUTCOMES:
clinical supervisor-rated communication skills performance | Baseline and immediately after completion of the intervention.
  Clinical supervisors evaluate interns' communication skills using the Gap-Kalamazoo Communication Skills Assessment Form (GKCSAF).
Patient-rated communication skills performance | Baseline and immediately after completion of the intervention.
  Patients evaluate interns' communication behavior using the Gap-Kalamazoo Communication Skills Assessment Form (GKCSAF).
Intern self-rated communication skills performance | Baseline and immediately after completion of the intervention.
  Interns complete a self-assessment using the Gap-Kalamazoo Communication Skills Assessment Form (GKCSAF).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Medical Hospital, Kaohsiung City, Niaosong Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No